CLINICAL TRIAL: NCT04464291
Title: An Epidemiological Survey to Establish the Spectrum of Circulating Serotypes of S. Pneumoniae, in Patients Older 18 Years: Healthy Carriage, Patients With Non-invasive and Invasive Pneumococcal Infections in the Russian Federation
Brief Title: An Epidemiological Survey to Establish the Spectrum of Circulating Serotypes of S. Pneumoniae, in Patients Older 18 Years
Acronym: SPECTRUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Interregional Association for Clinical Microbiology and Antimicrobial Chemotherapy (IACMAC) (Other)
Responsible Party: Principal Investigator, Roman Kozlov, President, The Interregional Association for Clinical Microbiology and Antimicrobial Chemotherapy (IACMAC)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IAC-SPECTRUM-2019
Record Dates: First submitted 2019-09-09; First posted 2020-07-09 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Pneumonia, Pneumococcal; Invasive Pneumococcal Disease; Acute Otitis Media
Keywords: Serotype; Streptococcus pneumoniae; Epidemiology; Antmicrobial resistance
MeSH Terms: conditions — Pneumonia, Pneumococcal; Otitis Media

STUDY DESIGN:
Intervention Model Description: Prospective Multicentre Microbiological study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with pneumococcal infection (Experimental): There will be assessing the prevalence of Streptococcus pneumoniae serotypes in the nasopharynx in healthy people; in middle ear liquid in patients with acute otitis media; in sputum and epithelial lining fluid in patients with community-acquired pneumonia; in spinal fluid in patients with invasive pneumococcal indection
  Interventions: Other: Detection of Streptococcus pneumoniae strains

INTERVENTIONS:
Other: Detection of Streptococcus pneumoniae strains — There will be detection of Streptococcus pneumoniae, serotype identification, susceptibility tests for penicillin, erythromycin, azithromycin, tetracycline, ciprofloxacin, levofloxacin, moxifloxacin and vancomycin

SUMMARY:
Pneumococcal conjugate vaccine was added to the National Immunization Program in Russia in 2014 which could affect the changes in pneumococcal serotypes in growing population. The purpose of this study is to determine the spectrum of serotypes of S. pneumoniae in patients older 18-years: in healthy carriage, in patients with non-invasive and invasive forms of pneumococcal infection. The patients will be divide into several groups: 18-64-years old, 65 years old and older, immunocompromised patients, immunocompetent patients with concomitant diseases and patients from restricted organized collectives.

This study is designed to meet the following objectives:

To estimate the spectrum of serotypes of S. pneumoniae in adult population in different regions of Russia.

DETAILED DESCRIPTION:
S. pneumoniae is a major cause of illness and death in children and adults worldwide. It includes 91 serotypes. The distribution of serotypes that cause disease varies by age, disease syndrome, disease severity, geographic region, and over time. Infants and young children are thought to be the main reservoir of this agent. From the colonized nasopharyngeal mucosa, pneumococci may spread by contiguous, non-invasive extension to other sites in the respiratory tract.

About 1.6 million cases of fatal pneumococcal disease occur worldwide annually, mostly in infants and the elderly.3 In addition, immunocompromised individuals of all ages, immunocompetent patients with concomitant diseases (chronic heart failure, broncho-obstructive syndrome, liquorrhea, ext.) are at increased risk.

Pneumococcal resistance to commonly used antimicrobials is a serious and increasing problem worldwide. Therefore vaccination is the most effective mechanism to reduce the incidence of pneumococcal infection in children and adult patients.

The effectiveness of pneumococcal vaccine is estimated by coverage of serotypes of S. pneumoniae. The distribution of the serotypes can be potentoinally changed because of the using of PCV in Russia.

Study design. Prospective Multicentre Microbiological study.

General informed consents are collected from patients at hospital admission. No additional informed consents will be collected for this study since the procedures of microbiological sample collection will be performed as a part of standard medical aid practices. Patient confidentiality will be retained at all times, and patient identifiers will not be included in the study. Collection of strains will be performed in patients, who meet inclusion criteria.

Inclusion Criteria

* Clinically relevant causative isolate - The isolate must meet the laboratory criteria of S. pneumoniae and be considered the "probable causative agent" of infection.
* Isolates from patients older 18-years with pneumococcal acute otitis media.
* Isolates from patients older 18-years with pneumococcal pneumonia
* Isolates from patients older 18-years with invasive pneumococcal diseases (meningitis, sepsis)
* Isolates from healthy carriage older 18-years Exclusion Criteria
* Isolates that have been collected and/or stored prior to June 1, 2018 or later than September 30, 2019.
* Duplicate isolates (same genus and species) obtained at any subsequent time from the same patient, regardless of susceptibility or phenotypic profile.
* Environmental samples (non patient-derived) or surveillance cultures taken for infection control purposes.
* Outside study group - Any isolate other than those defined by protocol.

Study procedures:

* collection of strains of S. pneumoniae and identification - the participating laboratory will collect, identify and store isolates and submit to reference laboratory of the Institute of Antimicrobial Chemotherapy of Smolensk State Medical University only clinical isolates that meet the study criteria as defined by protocol. Each isolate must be accompanied by a Organisms Report Form (ORF). The ORF contains information regarding the demographics of each isolate. Each investigative site will provide complete isolate identification using the laboratory's routine procedures.
* re-identification of strains of S. pneumoniae in the central laboratory (IAC, Smolensk) - at least, 500 consecutive non-duplicate strains of S. pneumoniae from healthy carriage and patients with non-invasive and invasive pneumococcal infections will be analyzed in centers from the following locations: Central region, North-Western region, Ural, Southern region, Siberia, Far-Eastern region. All the strains will be initially re-identified to the species level at the IAC laboratory using classic bacteriologic methods and MALDI Biotyper.
* susceptibility testing - susceptibility testing to penicillin, erythromycin, azithromycin, tetracycline, ciprofloxacin, levofloxacin, moxifloxacin and vancomycin will be determined by broth microdilution method. Interpretation will be done according to EUCAST/CLSI.
* serotyping (LATEX-TEST, Real-time PCR) - serotyping of S. pneumoniae will be performed using PNEUMOTEST-LATEX TEST and Real-Time PCR.
* data analysis
* reporting Strains collection: 01.06.2019 - 30.01.2020

Laboratory procedures:

1. Re-identification: till 31.10.2019
2. Antimicrobial susceptibility testing: till 01.06.2020
3. Serotyping: till 31.05.2020 Data analysis and reporting: till 28.02.2021 This is a non-interventional database study based on secondary use of data collected for other purposes. No administration of any therapeutic or prophylactic agent is required in this protocol. No reporting of individual adverse events to regulatory agencies is planned for this database study because there is no access to individual patient/subject records and it is not possible to assess the causality of individual cases. Pre-specified health outcomes of interest, including any that qualify as adverse events, will be summarized as part of any interim analysis (including safety analysis, if required) and in the final study report, which will be provided to regulatory agencies by the sponsor as required.

Any relevant safety information will be summarized in the appropriate Periodic Safety Update Report (PSUR)/Periodic Benefit Risk Evaluation Report (PBRER) and/or Development Safety Update Reports (DSUR) if required.

If an investigator elects to spontaneously report any suspected adverse reactions, they should be reported via fax to Merck AER Mailbox FAX #215-661-6229 (US), or toll-free fax 1-800-547-5552 (ex-US and US availability), in English using an AE form (attached) for reporting to worldwide regulatory agencies as appropriate

ELIGIBILITY:
Inclusion Criteria:

1. Clinically relevant causative isolate - The isolate must meet the laboratory criteria of S. pneumoniae and be considered the "probable causative agent" of infection.
2. Isolates from patients older 18-years with pneumococcal acute otitis media
3. Isolates from patients older 18-years with pneumococcal pneumonia
4. Isolates from patients older 18-years with invasive pneumococcal diseases (meningitis, sepsis)
5. Isolates from healthy carriage older 18-years

Exclusion Criteria:

1. Isolates that have been collected and/or stored prior to June 1, 2018 or later than September 30, 2019.
2. Duplicate isolates (same genus and species) obtained at any subsequent time from the same patient, regardless of susceptibility or phenotypic profile.
3. Environmental samples (non patient-derived) or surveillance cultures taken for infection control purposes.
4. Outside study group - Any isolate other than those defined by the protocol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of pneumococcal infection in the Russian Federation, caused by different serotypes of Streptococcus pneumoniae | 1 year
  The incidence will be detected with descriptive statistics

SECONDARY OUTCOMES:
Incidence of antimicrobial resistance of serotypes of Streptococcus pneumoniae | 1 year
  Detection of antimicrobial resistance to penicillin, erythromycin, azithromycin, tetracycline, ciprofloxacin, levofloxacin, moxifloxacin and vancomycin will be detected with descriptive statistics

CONTACTS AND LOCATIONS:
Locations (1):
- The Interregional Association for Clinical Microbiology and Antimicrobial Chemotherapy, Smolensk, Russia

IPD SHARING:
Plan to Share IPD: No